CLINICAL TRIAL: NCT04046991
Title: Treating Primary Progressive Aphasia (PPA) and Elucidating Neurodegeneration in the Language Network Using Transcranial Direct Current Stimulation (tDCS)
Brief Title: Treating Primary Progressive Aphasia (PPA) Using High-definition tDCS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 834650
Record Dates: First submitted 2019-07-12; First posted 2019-08-06 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Primary Progressive Aphasia
Keywords: non-invasive brain stimulation; transcranial direct current stimulation (tDCS); aphasia
MeSH Terms: conditions — Aphasia, Primary Progressive; Aphasia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- HD-tDCS+mCILT (Active Comparator): Participants will undergo 10 daily sessions (Monday-Friday, x2 weeks) of HD-tDCS for 20 minutes using a montage in which a central electrode (1.5mA) is placed over the left frontotemporal area and four surrounding cathodes (.375mA each). Subjects will participate in a modified constraint-induced language therapy.
  Interventions: Device: high-definition transcranial direct current stimulation; Behavioral: modified constraint-induced language therapy
- Sham+mCILT (Sham Comparator): Participants will undergo 10 daily sessions (Monday-Friday, x2 weeks) of sham for 20 minutes using a montage in which a central electrode is placed over the left frontotemporal area and four surrounding cathodes. Subjects will participate in a modified constraint-induced language therapy,
  Interventions: Device: high-definition transcranial direct current stimulation; Behavioral: modified constraint-induced language therapy

INTERVENTIONS:
Device: high-definition transcranial direct current stimulation — High definition transcranial direct current stimulation (HD-tDCS) involves the application of low-intensity current through electrodes placed on the scalp. It is believed to elicit brain effects by producing incremental shifts in the resting membrane potential of large numbers of neurons, which alters neuronal firing rates and thus modulates patterns of brain activity in potentially behaviorally-relevant ways. HD-tDCS differs from conventional transcranial direct current stimulation (tDCS) because it employed smaller electrodes configured in such a way as to deliver more focal stimulation of the brain.
Behavioral: modified constraint-induced language therapy — Modified constraint-induced language therapy (mCILT) is a behavioral language therapy that invokes use-dependent learning in communicative interactions by requiring spoken output and restricting use of alternative forms of communication, such as gestures, as a substitute for spoken output. Other key elements of CILT include massed practice of goal-directed speech and shaping of desired responses by increasing response demands as participants improve. MCILT differs from traditional constraint-induced language therapy (CILT) in three ways: 1) it will be done as an individual therapy with the examiner in the role of a communication partner; 2) treatment will be delivered in short sessions (1 hour rather than a more typical 3-4 hour session); 3) targeting nouns + semantically related verbs to generate noun + verb phrases in treatment, a modification that may be better suited to addressing syntactic structure.

SUMMARY:
This is a double-blind, sham-controlled, crossover study in which subjects with the non-fluent/agrammatic and logopenic variants of primary progressive aphasia (naPPA and lvPPA, respectively) will undergo language testing and structural and functional brain imaging before and after receiving 10 semi-consecutive daily sessions of real or sham high-definition transcranial direct current stimulation (HD-tDCS) paired with modified constraint-induced language therapy (mCILT). Language testing and brain imaging will be repeated immediately after completion of and 3 months following completion of treatment. The 3-month follow-up will be the primary endpoint. The investigators will examine changes in language performance induced by HD-tDCS + mCILT compared to sham HD-tDCS + mCILT. The investigators will also use network science to analyze brain imaging (fMRI) data to identify network properties associated with baseline PPA severity and tDCS-induced changes in performance. This study will combine knowledge gained from our behavioral, imaging, and network data in order to determine the relative degrees to which these properties predict whether persons with PPA will respond to intervention.

DETAILED DESCRIPTION:
The central framework for the project is a double-blind, sham-controlled, crossover study in which subjects with the non-fluent/agrammatic and logopenic variants of primary progressive aphasia (naPPA and lvPPA, respectively) will undergo language testing and structural and functional brain imaging before and after receiving 10 semi-consecutive daily sessions of real or sham high definition transcranial direct current stimulation (HD-tDCS) paired with modified constraint-induced language therapy (mCILT). Language testing and brain imaging will be repeated immediately after completion of and 3 months following completion of treatment.

Subjects with naPPA and lvPPA will be randomized to one of two study arms: HD-tDCS+mCILT or sham stimulation+mCILT paired with pre- and post-stimulation imaging and behavioral measures. Equal numbers of subjects with naPPA and lvPPA will be randomized to the HD-tDCS + mCILT and sham + mCILT study arms. The study is double-blinded, in that neither the subject nor the study personnel administering HD-tDCS or sham stimulation will know which arm of the study the subject has been randomized into. Study coordinators will administer HD-tDCS by entering a pre-determined code that has been programmed into the device by another member of the study team. Data will be digitally audio-recorded and analyzed off-line, such that study team members performing data coding and analysis will likewise be blinded to the treatment condition of each subject.

Subject participation in this protocol will occur during 27 planned visits that will span approximately 8 months. The events of the study visits are described below:

VISIT 1:

a Informed consent and screening b. Baseline language assessment #1 c. Baseline MRI scanning

VISIT 2:

Baseline language assessment #2

VISITS 3-11:

HD-tDCS+mCILT OR sham stimulation+mCILT, depending on the study arm to which they had been randomized.

VISIT 12:

1. Final session of HD-tDCS+mCILT or sham stimulation+mCILT
2. Follow-up language assessment
3. Follow-up MRI

VISIT 13:

6-Week follow-up language assessment

VISIT 14:

1. 12-week follow-up language assessment
2. 12-week follow-up MRI

**CROSSOVER**

VISIT 15:

Crossover baseline language assessment #2

VISITS 16-24:

HD-tDCS+mCILT or sham stimulation+mCILT

VISIT 25:

1. 10th session of HD-tDCS+mCILT or sham stimulation+mCILT
2. Follow-up language assessment
3. Follow-up MRI

VISIT 26:

6 Week follow-up language assessment:

VISIT 27:

1. 12-week follow-up language assessment
2. 12-week follow-up MRI

ELIGIBILITY:
Inclusion Criteria:

1. Presence of aphasia attributable to nonfluent agrammatic PPA (naPPA) or logopenic variant PPA (lvPPA)
2. High school education (or more)
3. Must be able to understand the nature of the study, and give informed consent
4. Native English speaker

Exclusion Criteria:

* Presence of additional neurological illness such as stroke or traumatic brain injury
* Diagnosis of epilepsy or reoccurening seizures
* Pacemaker or ICDs
* Craniotomy or skull breech
* Small vessel disease

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Western Aphasia Battery Aphasia Quotient (WAB-AQ) | Baseline, 2 weeks, 6 weeks, 12 weeks, 14 weeks, 18 weeks, 24 weeks
  The primary outcome measure will be the change in score on the WAB-AQ, a score assessing overall aphasia recovery. Scores can range from 0-100. 0-25 is very severe, 26-50 is severe, 51-75 is moderate, and 76-above is mild. A score of 93 or higher is considered recovered.

CONTACTS AND LOCATIONS:
Overall Officials: Roy H Hamilton, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States